CLINICAL TRIAL: NCT03280940
Title: Impact of Different Integrase Inhibitor Based Regimen on Markers of Inflammation and Immune Activation Among HIV naïve Patient During the First Year of Effective First-line Combination
Brief Title: Impact of Different Integrase Inhibitor Based Regimen on Immune Activation Among HIV naïve Patient (INTATTI)
Acronym: INTATTI
Status: Completed | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, EUGENIA QUIROS ROLDAN, Prof., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: INTATTI
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: HIV Infections
Keywords: Inflammation; Immune activation; Integrase Inhibitors; Naive patients
MeSH Terms: conditions — HIV Infections; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum (Biospecimen retained as a normal clinical practice)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Dolutegravir treatment group: Naïve patients having documented HIV-1 infection and starting their first antiretroviral treatment with a dolutegravir containing regimen
- Raltegravir treatment group: Naïve patients having documented HIV-1 infection and starting their first antiretroviral treatment with a raltegravir containing regimen
- Elvitegravir treatment group: Naïve patients having documented HIV-1 infection and starting their first antiretroviral treatment with a elvitegravir containing regimen
- Protease inhibitors treatment group: Naïve patients having documented HIV-1 infection and starting their first antiretroviral treatment with a protease inhibitors containing regimen

SUMMARY:
Low viral replication persistence and immune activation remain important therapeutic challenge in the new HAART era. They are associated with more rapid disease progression, increased risk of mortality and non-AIDS defining events. Soluble biomarkers are a convenient way of assessing immune activation and inﬂammation in HIV-infected patients receiving effective treatment. There are limited data describing the different effects of currently recommended antiretroviral regimens on immune activation and inﬂammation during HIV infection. Several studies have shown that raltegravir (the first approved drug from integrase inhibitor class) seems to have more impact on decreasing systemic inflammation compared with other drug classes. Integrase inhibitors may decrease inflammation and immune activation more than other antiretroviral drugs, because they are more lipid friendly and may concentrate better in enterocytes. The aim of this observational study is to compare the impact of different integrase inhibitor based regimen on changes in markers of inflammation (Il-2, IL-6, sTNFR-1, sCD14, sCD163, sICAM, hsRCP , sVCAM, LPS, D-dimer) during the first year of effective first-line combination. This is a 48-week observational retrospective study, to compare the change in infiammatory markers between naïve patients who start INI based regimen. Participants will be recruited from the HIV outpatient clinic. The study compare the impact of commonly used first-line antiretroviral drugs on soluble markers of inflammation and immune activation. The study is conducted on treatment-naive HIV-infected patients who experience a rapid and persistent virological response and that do not switch their initial regimen for at least 1 years. The analyses will be adjusted for baseline characteristics that might influence the choice of cART regimen or affect biomarker levels, such as age, smoking status, CD4 cell count, plasma HIV-1 viral load. Investigators enroll patients with a rapid and persistent virological response and that do not experience any blips. Cryopreserved plasma sample are obtained at baseline and at month 6 and 12 after treatment starting. Two NRTI backbone combinations (TDF/FTC vs ABC/3TC) and three third agents (RAL vs ELV vs DTG) will be compared in a factorial design. The results will be expressed as the estimated percentage difference between the mean fold changes observed with a given drug, using TDF/FTC and RAL as the reference groups for the comparison.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND Combination antiretroviral therapy (cART) controls HIV-1 plasma viral load in most patients, leading to a reduction in morbidity and mortality [Egger M, BMJ 1997; Detels R, JAMA 1998].

Despite efficient treatment persistent low-level viral replication and immune activation remain an important therapeutic challenge. Immune activation is associated with more rapid disease progression and with less efﬁcient CD4+ cell recovery during cART [Hunt PW, J Infect Dis 2003; Lederman MM, J Infect Dis 2011], while plasma biomarkers of inﬂammation have been linked to a risk of mortality and non-AIDS-deﬁning events such as cardiovascular disease and non-AIDS-deﬁning cancers [Kuller LH, PLoS Med. 2008; Ipp H, Clin Chim Acta. 2013].

A potential link between HIV-associated inﬂammation and disease progression and mortality was shown for the first time in a randomized clinical trial of continuous versus intermittent antiretroviral therapy (the Strategies for Management of Antiretroviral Therapy study - SMART study) [Neuhaus J, J Infect Dis 2010]. In this study HIV-infected persons were randomized to continuous antiretroviral therapy (ART) or CD4- T cell count- driven ART. Subjects randomized to the second arm had a higher risk of morbidity and mortality. ART interruption resulted in a rapid increase in inﬂammation- and coagulation-associated biomarkers that were associated with increased risks of death, AIDS, and cardiovascular disease (CVD).

Further studies have confirmed that HIV-infected individuals have elevated levels of inﬂammatory and cellular activation markers and suppression of viral replication by ART decreases, but does not normalize those markers [Regidor DL, AIDS 2011; Widney DP, J Interferon Cytokine Res 2005; Kaplan RC, J Acquir Immune Deficiency Syndr 2012].

Soluble biomarkers are a convenient way of assessing immune activation and inﬂammation in HIV-infected patients receiving cART. Interleukin-6 (IL-6) is a biomarker of inﬂammation and was found to be associated with all-cause mortality and cardiovascular diseases in the SMART study [Neuhaus J, J Infect Dis 2010]. Interferon-γ-inducible protein-10 (IP-10) and monokine induced by interferon-γ (MIG) are two chemokines produced by different cells and target lymphocytes, particularly activated T cells. Elevated plasma IP-10 levels during the primary phase of HIV-1 infection were predictive of earlier decline in the CD4 cell count in a recent study [Liovat AS, PLOS One 2012; Jiao Y, Viral Immunology 2012; N. Noel, IAS 2013]. Soluble CD14 (sCD14) is a marker of monocyte activation that binds to lipopolysaccharides in plasma. Plasma levels of sCD14 are an independent predictor of mortality among HIV-infected patients [D Sandler et al , JID 2011; E Krastinova, J Infect Dis. 2015] .

There are limited data describing the differential effects of currently recommended antiretroviral regimens on immune activation and inﬂammation during HIV infection. As long as viral suppression remains the goal of HIV treatment, choosing ART with the least long -term toxicity and highest beneﬁt is of great priority in the management of this chronic illness.

Understanding how different ART regimens reduce chronic immune activation and inflammation in treated HIV-infected patients is an ongoing interesting research.

Several studies have shown that raltegravir (the first approved drug from integrase inhibitor class) seems to have more impact on decreasing systemic inflammation compared with drugs from protease inhibitor or non-nucleside transcriptase inhibitor classes [Asmuth DM, AIDS 2012; Massanella M, AIDS 2012; Asmuth DM, AIDS 2014], both in naïve or treated-virologically suppresed patients [Gupta SK, J Acquir Immune Defic Syndr. 2013; Lake JE, HIV Medicine 2014].

It is plausible that drugs from integrase inhibitor class may decrease inflammation and immune activation more than other antiretroviral classes, because they are more lipid friendly and may concentrate better in enterocytes [ Martinez E, AIDS 2010] [Patterson KB, AIDS 2013].

The aim of this observational study is to compare the impact of different INI based regimen on changes in markers of inflammation (Il-2, IL-6, sTNFR-1, sCD14, sCD163, sICAM, hsRCP , sVCAM, LPS, D-dimer) during the first year of effective first-line combination.

OBJECTIVES The primary objective is to evaluate the changes in markers of inflammation (Il-2, IL-6, sTNFR-1, sCD14, sCD163, sICAM, hsRCP , sVCAM, LPS, D-dimer) in patients who receive first line INI-based therapy.

METHODS This is a 48-week observational retrospective study, to compare the change in infiammatory markers between naïve patients who start INI based regimen. Participants will be recruited from the HIV outpatient clinic.

STUDY DESIGN The study will compare the impact of commonly used first-line antiretroviral drugs on soluble markers of inflammation and immune activation. In order to avoid the influence of previous ARV exposure, active viral replication and treatment switches, the analysis is limited to a homogenous group of treatment-naive HIV-infected patients who experience a rapid and persistent virological response and remain on their initial regimen for 1 years. The evaluation of biomarkers of inflammation is not a part of rourtine analysis, so investigators will enrolled patients who have plasma samples stored before ART initiation, 6 month and 1 year later.

The analyses will be adjusted for baseline characteristics that might influence the choice of cART regimen or affect biomarker levels, such as age, smoking status, CD4 cell count, plasma HIV-1 viral load. Patients who had a rapid and persistent virological response (defined by a plasma HIV-1 viral load (VL) below 400 copies/mL at 6 months and below 50 copies/mL at 12 months), with no values above 1000 copies/ml between month 6 and month 12 are enrolled in this study, in order to control potential causes of inflammation/activation due to persistent plasma viral replication Inclusion criteria

1) Naïve patients having documented HIV-1 infection, of age 18 years and older Exclusion criteria

1. Patients with diagnosed CVD, diabetes, uncontrolled hypertension (screening systolic blood pressure >160 mm Hg or diastolic pressure >90 mm Hg),
2. other systemic inflammatory disease (hepatitis B or C coinfection was allowed)
3. estimated creatinine clearance <70 mL/min;
4. HIV-1 RNA level of <1000 copies/mL,
5. prior ART use
6. estimated glomerular filtration rate (eGFR) of <70 mL/min by the Cockcroft-Gault equation
7. liver transaminase levels <5 times the upper limit of normal
8. absolute neutrophil count of <1000 neutrophils/mm3
9. platelet count of ≥50 000 platelets/mm3,
10. hemoglobin level of ≥8.5 g/dL,
11. use of lipid-lowering drugs
12. life expectancy of ≥1 year from the time of enrollment
13. AIDS-defining conditions diagnosed within 30 days
14. active infection or malignancy
15. current alcohol or substance use judged to potentially interfere with study compliance Markers of Inflammation and Immune Activation Cryopreserved plasma sample were obtained at baseline (prior to ART initiation) and at month 6 and 12 after treatment starting from 30 patients participating at MASTER (Management of Standardized Evaluation of Retroviral HIV Infection) group, an ongoing prospective multicentre cohort that includes the major Italian clinical centres involved in HIV infection care.

Thawed samples will stained for this circulating inflammatory markers [high sensitivity C-reactive protein (hsCRP), serum interleukin-6 (IL-6), interleukin-2 (IL-2), soluble tumor necrosis factor-[alpha] receptors I and II (sTNFRI and sTNFRII), endothelial markers (soluble vascular cell adhesion molecule-1,), markers of monocyte/macrophage activation [soluble CD14 (sCD14), soluble CD163 (sCD163)], D-dimer.

Statistical analysis The aim of this exploratory study is to evaluate the effect of a new integrase inhibitor on serum level of inflammatory markers.

Two NRTI backbone combinations (TDF/FTC vs ABC/3TC) and three third agents (RAL vs ELV vs DTG) will be compared in a factorial design. Baseline characteristics will be compared between treatment groups by using the Wilcoxon and chi-squared tests in order to identify variables associated with the choice of treatment. Because the marker values isn't normally distributed, they will be log e-transformed for analysis. For each marker, changes between D0, M6 and M12 (mean fold change) will be expressed as the geometric mean of their ratio after log-e transformation. A paired one-sample t test will be used to identify significant differences in the overall changes in each marker. Linear regression models will be used to investigate the impact of the different NRTI backbones and the different third agents on the biomarker changes. The results will be expressed as the estimated percentage difference between the mean fold changes observed with a given drug, using TDF/FTC and RAL as the reference groups for the comparison. Relationships between baseline covariables and changes in each biomarker will be examined in univariable linear regression models. These covariables will be sex, age, body mass index, smoking status, prior AIDS-defining events, and the pre-ART CD4 cell count and viral load. Baseline covariables associated with changes in at least one biomarker (p < 0.10) and viral blips above 50 copies/ml between M6 and M12 will be retained in all multivariable linear regression models in order to control for factors that might have influenced the choice of cART regimen or affected biomarker levels. Age and smoking status will be included in the multivariable model since these variables are known to influence marker levels. Interaction terms between the NRTI backbone and the third agent will be tested for each marker. Sensitivity analyses will conduct. Statistical analyses will run on STATA 12 software, and p values <0.05 were considered statistically significant.

Ethics This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and will be consistent with Good Clinical Practice (GCP) and applicable regulatory requirements.

The study will be conducted in compliance with the protocol. The protocol and any amendments and the patient informed consent will receive Ethics Committee (EC) approval/favourable opinion prior to initiation of the study.

Freely given written informed consent must be obtained from every patient or their legally acceptable representative prior to clinical trial participation, including informed consent for any screening procedures conducted to establish patient eligibility for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Naïve patients having documented HIV-1 infection, of age 18 years and older

Exclusion Criteria:

1. Patients with diagnosed CVD, diabetes, uncontrolled hypertension (screening systolic blood pressure >160 mm Hg or diastolic pressure >90 mm Hg),
2. Other systemic inflammatory disease (hepatitis B or C coinfection was allowed)
3. Estimated creatinine clearance <70 mL/min;
4. HIV-1 RNA level of <1000 copies/mL,
5. Prior ART use
6. Estimated glomerular filtration rate (eGFR) of <70 mL/min by the Cockcroft-Gault equation
7. Liver transaminase levels <5 times the upper limit of normal
8. Absolute neutrophil count of <1000 neutrophils/mm3
9. Platelet count of ≥50 000 platelets/mm3
10. Hemoglobin level of ≥8.5 g/dL
11. Use of lipid-lowering drugs
12. Life expectancy of ≥1 year from the time of enrollment
13. AIDS-defining conditions diagnosed within 30 days
14. Active infection or malignancy
15. Current alcohol or substance use judged to potentially interfere with study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naive HIV-infected patients followed at University Division of Infectious and Tropical Diseases, University of Brescia (Italy) who experience a rapid and persistent virological response and remain on their initial regimen for 1 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Inflammation outcomes 48 week | 48 week
  Evaluate the changes from baseline to week 48 in level of markers of inflammation (IL-2, IL-6, sTNFR-1, sCD14, sCD163, sICAM, hsRCP , sVCAM, LPS, D-dimer) in patients who receive first line antiretroviral therapy

SECONDARY OUTCOMES:
Inflammation outcomes 24 week | 24 week
  Evaluate the changes from baseline to week 24 in level of markers of inflammation (IL-2, IL-6, sTNFR-1, sCD14, sCD163, sICAM, hsRCP , sVCAM, LPS, D-dimer) in patients who receive first line antiretroviral therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Quiros Roldan, Prof, Principal Investigator — AO Spedali Civili di Brescia
Locations (1):
- AO Spedali Civili di Brescia, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: No